CLINICAL TRIAL: NCT06064084
Title: Incretin Effect in Patients With Psoriasis
Brief Title: Incretin Effect in Patients With Psoriasis and Controls
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, MD, University Hospital, Gentofte, Copenhagen
Other Study IDs: 11031999
Record Dates: First submitted 2023-09-14; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriasis
  Interventions: Diagnostic Test: Oral glucose tolerance test; Other: Intravenous isoglycaemic glucose clamp; Other: Liquid Mixed meal test
- Control: Age, Sex and BMI matched
  Interventions: Diagnostic Test: Oral glucose tolerance test; Other: Intravenous isoglycaemic glucose clamp; Other: Liquid Mixed meal test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — Oral glucose tolerance test 50g
Other: Intravenous isoglycaemic glucose clamp — Intravenous isoglycaemic glucose clamp
Other: Liquid Mixed meal test — Liquid Mixed meal test 520 kcal

SUMMARY:
To investigate the incretin effect and postprandial incretin responses in plasma in patients with psoriasis

ELIGIBILITY:
Inclusion Criteria:

no diabetes BMI < 27 kg/m^2 normal Glucose tolerance test at screening normal fasting plasma glucose no islet auto antibodies no hormonel contraception informed consent psoriasis vulgaris (PASI>8) (case not controls)

Exclusion Criteria:

other chronic inflammtory skin disease other chronic inflammatory disease pregnancy psychiatric illness

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Cases with psoriasis vulgaris (PASI>8) Controls with no existing skin disease. Matched for Age, BMI and Sex
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-09-11 (Actual); Primary Completion 2015-09-11 (Actual); Study Completion 2015-09-11 (Actual)

PRIMARY OUTCOMES:
Incretin effect measured with Beta-cell secretory response | 0-180 minutes
  Incretineffect (%) = 100 % × (Beta-cell Secretory Response (OGTT) - Beta-cell Secretory Response (IIGI)) / Beta-cell Secretory Response (OGTT)

SECONDARY OUTCOMES:
Insulin sensitivity measures | 0-180 minutes
  Matsudas insulin sensitivity index: (10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT))
Concentration of Glucose-independent insulinotropic polypeptide | 0-180 minutes
  Evaluted as Area Under the Curve
Concentration of Glucagon-like peptide 1 | 0-180 minuntes
  Evaluated as Area Under the Curve
Concentration of Glucagon | 0-180 minutes
  Evaluated as Area Under the Curve
Concentration of Insulin | 0-180 minutes
  Evaluated as Area Under the Curve

REFERENCES:
- [Derived] Lauritsen JV, Bergmann N, Junker AE, Gyldenlove M, Skov L, Gluud LL, Hartmann B, Holst JJ, Vilsboll T, Knop FK. Oral glucose has little or no effect on appetite and satiety sensations despite a significant gastrointestinal response. Eur J Endocrinol. 2023 Dec 6;189(6):619-626. doi: 10.1093/ejendo/lvad161. PMID 38035766